CLINICAL TRIAL: NCT01893931
Title: Discharge Planning for Older Adults in the Emergency Department: Use of a Brief Phone Call After Discharge to Decrease Return Visits to the Emergency Department and Re-admissions to the Hospital
Brief Title: Use of a Brief Phone Call After ED Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The William R. Kenan, Jr. Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-1278
Record Dates: First submitted 2013-06-24; First posted 2013-07-09 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Discharge Planning; Emergency Medicine; Geriatrics; Patient Readmission
Keywords: Geriatrics; Emergency Medicine; Care Transitions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Satisfaction Survey (Placebo Comparator): Within 1-3 days after ED discharge, patients will be called by a nurse to complete a brief satisfaction survey.
  Interventions: Behavioral: Placebo Comparator
- ED Discharge and Medication Call (Active Comparator): Within 1-3 days after ED discharge, patients will receive a follow up phone call from a nurse to review discharge instructions, review medication instructions, and provide any necessary patient navigation.
  Interventions: Behavioral: ED Discharge & Medication Call

INTERVENTIONS:
Behavioral: ED Discharge & Medication Call — Patients will receive a follow up phone call from a nurse to review discharge instructions and provide any necessary patient navigation.
  Arms: ED Discharge and Medication Call
Behavioral: Placebo Comparator
  Arms: Satisfaction Survey

SUMMARY:
The purpose of this study is to determine whether a phone call from a nurse within 1-3 days after discharge from the Emergency Department (ED) decreases return visits to the ED/ hospital admissions/ death (combined outcome) in patients age 65 and above. As secondary outcomes, time to follow up appointment with physician and economic impact of this intervention will be assessed.

Patients 65 years of age and older will be randomized following discharge from the ED into one of two groups. Group 1(Intervention) will receive a phone call collecting information about understanding of ED discharge instructions and guiding patient through the discharge instructions, and Group 2 (Placebo) will receive a follow up phone call for a satisfaction survey.

We hypothesize return visits to the ED and readmission to the hospital will decrease as a result of the nurse phone call intervention.

DETAILED DESCRIPTION:
Procedures: All patients age 65 and above will be randomized to one of two groups within 1-3 days after discharge from the UNC ED: 1) Interventional follow-up phone call; or 2) Placebo phone call, implementing only a satisfaction survey.

The intervention phone call will ask whether patients have obtained the newly prescribed medicines, ask if the patient understands the instructions for taking the medicines and inquire if a patient has made an appointment with his/her personal physician. The caller will attempt to answer questions about the medicines, and encourage patients to take the medicines as directed. The caller will also encourage the patients to follow-up with their own physician in a timely manner and offer to help with setting up follow up appointments if needed.

Subsequently, 30-35 days after ED discharge, all patients will receive a phone call to evaluate rates of compliance with medicines and scheduling follow-up appointments. All calls will be made by trained nurses.

Using an α 0.05 and β 0.80 we will need to enroll 2235 patients to detect a decrease in ED return visits/re-admission/ death of 6%. There will be one interim analysis 1 year into the two year planned study.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 65 and above discharged from the ED
* English speaking

Exclusion Criteria:

* Younger than 65 years of age
* Unable to pass 6-item memory screener
* Lives in skilled nursing facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2003 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Time to the first occurrence of hospital readmission, emergency department visit, or death. | 0-35 days
  Measured by (1) Self-report via a phone call to the patient or care giver up to 35 days post-discharge, and (2) Utilization of existing medical records.

SECONDARY OUTCOMES:
Time elapsed from initial emergency department visit to Physician follow up | 0-35 Days
Patient satisfaction as reported by phone survey | 0-35 Days

CONTACTS AND LOCATIONS:
Overall Officials: John S Kizer, M.D., Principal Investigator — University of North Carolina, Chapel Hill; Kevin Biese, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biese KJ, Busby-Whitehead J, Cai J, Stearns SC, Roberts E, Mihas P, Emmett D, Zhou Q, Farmer F, Kizer JS. Telephone Follow-Up for Older Adults Discharged to Home from the Emergency Department: A Pragmatic Randomized Controlled Trial. J Am Geriatr Soc. 2018 Mar;66(3):452-458. doi: 10.1111/jgs.15142. Epub 2017 Dec 22. PMID 29272029